CLINICAL TRIAL: NCT01563159
Title: Assessing the Rotavirus Positive Test Results in 11 Hospitals in Belgium From 2005 to 2013: the RotaBIS Study (Rotavirus Belgian Impact Study)
Brief Title: Number of Rotavirus (RV) Related Hospitalizations in Belgium - Season 2010-2011
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116312
Record Dates: First submitted 2012-03-01; First posted 2012-03-26 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Infections, Rotavirus
Keywords: Belgium; hospitals; Rotavirus
MeSH Terms: conditions — Rotavirus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: All children ≤ 5 years old with a rotavirus detection test (inpatient and ambulatory tests) performed during the period of June the 1st 2010 and May the 31st 2011.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Each participating centre will be requested to generate a coded list of all stool samples taken during the study period (June 1st 2010- May 31st 2011) and analysed for rotavirus, in children aged ≤5 years.

SUMMARY:
This study aims to confirm the statistically significant decline in rotavirus related and in acute gastro-enteritis (AGE) related hospital admissions that was observed in 11 participating hospitals, after the introduction of RV vaccines in Belgium in 2006.

DETAILED DESCRIPTION:
This retrospective study will use anonymised data, extracted from hospital databases during the period of the 1st of June 2010 until the 31st of May 2011. IMS Health sales data will be used to provide rotavirus vaccine coverage estimates (Rotarix and Rotateq) for the Belgian population during the study period. Any additional source of vaccine coverage status describing rotavirus vaccine uptake in the study population will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Child aged ≤5 years;
* A stool sample has been provided for a rotavirus detection test during the study period;
* Laboratory test result of rotavirus is available.

Exclusion Criteria:

Not applicable.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged ≤5 years undergoing a RV detection test across 11 participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Absolute number of rotavirus related hospitalisations in children up to five years old. | During the study period (from June 1st 2010 to May 31st 2011, i.e. up to 1 year)

SECONDARY OUTCOMES:
Proportion of rotavirus positive tests on the total number of rota detection tests | During the study period (from June 1st 2010 to May 31st 2011, i.e. up to 1 year)
  Total number of rota detection tests and number of rotavirus positive tests of the study year will be determined by age-group of 1-year, gender, time of the event, vaccine coverage status.
The duration of rota-related hospitalisation for community acquired and nosocomial infection. | During the study period (from June 1st 2010 to May 31st 2011, i.e. up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Standaert B, Strens D, Pereira P, Benninghoff B, Raes M. Lessons Learned from Long-Term Assessment of Rotavirus Vaccination in a High-Income Country: The Case of the Rotavirus Vaccine Belgium Impact Study (RotaBIS). Infect Dis Ther. 2020 Dec;9(4):967-980. doi: 10.1007/s40121-020-00345-y. Epub 2020 Oct 6. PMID 33025558